CLINICAL TRIAL: NCT00542412
Title: Care (Canadian ALS Riluzole Evaluation) Multicentre Phase IV Comparative Study of the Effects of Riluzole 50mg Bid on the Survival of ALS Subjects Compared to Historical Controls
Brief Title: CARE Canadian ALS Riluzole Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIL_CA1_401
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Riluzole

SUMMARY:
Evaluate the efficacy of riluzole 50-mg bid defined by comparing the percentage of riluzole-treated subjects who experienced death, permanently assisted ventilation (PAV) or tracheostomy, to a group of recent historical controls for the treatment of amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS confirmed by the following definition:

  (a)"Probable" or "Definite" Amyotrophic Lateral Sclerosis (ALS) according to the El Escorial criteria(b)"Peripheral" onset form (limb involvement) or a "Bulbar" form of ALS with a duration of five years, based on inquiry for the earliest symptoms of the disease
* A subject who simultaneously presents with bulbar and peripheral signs at onset of ALS disease should be stratified to the bulbar onset group. The neurologic progression of such subjects matches that of the bulbar onset ALS subjects.
* Pulmonary Function: forced vital capacity (FVC) must be 3 60% at study entry.
* Females of childbearing potential must be documented to be using acceptable birth control methods such as an IUD or oral contraceptives.

Exclusion Criteria:

* Previous treatment with riluzole
* Tracheostomy, or expected to undergo a tracheostomy within two months after study inclusion
* Signs of clinical dementia and/or major psychiatric disorders
* Serious concomitant disease or handicap likely to interfere with the subject's assessments or impact on the subject's survival
* A multiple conduction block has been shown on nerve conduction studies by electromyogram

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2001-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the time to the occurrence of an ALS-related event (PAV, tracheostomy or ALS-related death)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent-Didier Jacobs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Laval, Quebec, Canada